CLINICAL TRIAL: NCT03812068
Title: The Effectiveness of a Parent-mediated Developmental Behavioral Intervention for Children With Autism Spectrum Disorder and Developmental Delay: A Randomized Controlled Trial
Brief Title: Parent-mediated Developmental Behavioral Intervention
Acronym: PDBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201809001RINC
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-10

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; Early intervention; Development
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-distance developmental behavioral intervention (Experimental): Long-distance learning program combined parent-mediated developmental behavioral intervention
  Interventions: Behavioral: Long-distance developmental behavioral intervention
- Developmental behavioral intervention (Active Comparator): only parent-mediated developmental behavioral intervention
  Interventions: Behavioral: Developmental behavioral intervention

INTERVENTIONS:
Behavioral: Long-distance developmental behavioral intervention — Long-distance learning program combined parent-mediated developmental behavioral intervention
  Arms: Long-distance developmental behavioral intervention
Behavioral: Developmental behavioral intervention — Parent-mediated developmental behavioral intervention
  Arms: Developmental behavioral intervention

SUMMARY:
This study explores the effectiveness of two intervention programs: "Long-distance developmental behavioral intervention" and "developmental behavioral interventions" for children with autism spectrum disorder or multiple developmental delays.

ELIGIBILITY:
Inclusion Criteria:

* Child's age between 30-84 months old.
* Children have a diagnosis of autism spectrum disorder or multiple developmental delays.
* Children without physical disabilities or major health problems, such as congenital limb defects.
* One of the fathers or mothers involved in the study shall be the primary caregiver of the child.
* The father or mother participating in the study has at least 9 education years and can read and understand Chinese.
* The father or mother participating in the study is willing to allow the child to undergo a comprehensive development assessment and is willing to video during the training process.

Exclusion Criteria:

* Absence of chromosome abnormalities, congenital anomalies, and major neurological or sensory impairments or disorders (e.g., cerebral palsy, microcephalus, macrocephalus, severe brain damage, uncorrected vision, or hearing loss).

Min Age: 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
The Autism Diagnostic Observation Schedule | 3 months
  measurement of autism status and severity level
Child Behavior Checklist Ages 1.5-5 | 3 months
  measurement of child's behavioral syndrome and problems
Pediatric Evaluation of Disability Inventory | 3 months
  measurement of child's daily living function
Mullen Scale of Early Learning | 3 months
  measurement of child's cognitive and motor development
Movement Assessment Battery for Children | 3 months
  measurement of child's motor coordination
3D Gait Assessment Foot-worn Inertial Sensor | 3 months
  measurement of gait performance
Peabody Developmental Motor Scales, Second Edition | 3 months
  measurement of multiple fine and gross motor functions

SECONDARY OUTCOMES:
Parenting Stress Index | 3 months
  measurement of parenting stress for parents
Parenting Sense of Competence Scale | 3 months
  measurement of the parent's self-efficacy and satisfaction as being parents

CONTACTS AND LOCATIONS:
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided